CLINICAL TRIAL: NCT03527745
Title: Efficacy and Safety of Ascending Dosages of Albendazole Against T. Trichiura and Hookworm in Preschool- and School-aged Children and Adults: a Randomized Controlled Trial
Brief Title: Albendazole Dose Finding and Pharmacokinetics in Children and Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: Centre Suisse de Recherches Scientifiques en Cote d'Ivoire (Other)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Prof. Jennifer Keiser, PhD, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2018-05-03; First posted 2018-05-17 (Actual); Results first posted 2021-01-06 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Trichuriasis; Hookworm Infections
MeSH Terms: conditions — Trichuriasis; Hookworm Infections | interventions — Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 200 mg albendazole (Experimental): against T. trichiura in preschool-aged children or against hookworm infections in preschool-aged children, school-aged children and adults
  Interventions: Drug: Albendazole
- 400 mg albendazole (Experimental): against T. trichiura in preschool-aged children, school-aged children and adults or against hookworm infections in preschool-aged children, school-aged children and adults
  Interventions: Drug: Albendazole
- 600 mg albendazole (Experimental): against T. trichiura in preschool-aged children, school-aged children and adults or hookworm infections in preschool-aged children, school-aged children and adults
  Interventions: Drug: Albendazole
- 800 mg albendazole (Experimental): against T. trichiura in school-aged children and adults or against hookworm infections in school-aged children and adults
  Interventions: Drug: Albendazole
- Placebo (Placebo Comparator): against T. trichiura in preschool-aged children, school-aged children and adults or hookworm infections in preschool-aged children, school-aged children and adults
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albendazole — Single dose of albendazole (200mg, dependent on treatment cohort)
  Other Names: Zentel®
  Arms: 200 mg albendazole
Drug: Albendazole — Single dose of albendazole (400mg, dependent on treatment cohort)
  Other Names: Zentel®
  Arms: 400 mg albendazole
Drug: Albendazole — Single dose of albendazole (600mg, dependent on treatment cohort)
  Other Names: Zentel®
  Arms: 600 mg albendazole
Drug: Albendazole — Single dose of albendazole (800mg, dependent on treatment cohort)
  Other Names: Zentel®
  Arms: 800 mg albendazole
Drug: Placebo — Matching placebo tablets will be obtained from Fagron, Germany.
  Arms: Placebo

SUMMARY:
This study is a single-blind randomized clinical trial conducted in rural Côte d'Ivoire. This study aims at providing evidence on the dose-response of increasing oral albendazole dosages against whipworm (T. trichiura) and hookworm infections in preschoolers (2-5 years), school-aged children (6-12 years) and adults (≥ 21 years).

The primary objective is to determine cure rates (primary end point, i.e. conversion from being egg positive pre-treatment to egg negative post-treatment). Secondary objectives involve the determination of egg reduction rates (the reduction in the number of excreted eggs from baseline (prior to treatment) to follow-up) and the assessment of safety of ascending dosages of albendazole (secondary end points). In addition, key pharmacokinetic parameters will be determined from blood samples collected with a micro-sampling device (secondary end point).

DETAILED DESCRIPTION:
This study is a single-blind randomized clinical trial conducted in Côte d'Ivoire. This study aims at providing evidence on the efficacy and safety of ascending oral albendazole dosages in children and adults infected with T. trichiura and hookworm. In preschool-aged children (2-5 years) (i) 200 mg, (ii) 400 mg and (iii) 600 mg; in schoolchildren (6-12 years) and adults (≥ 21 years) (i) 200 mg (only for hookworm infections), (ii) 400 mg, (iii) 600 mg and (iv) 800 mg will be administered and efficacy, safety and pharmacokinetic parameters will be assessed.

The primary objective is to determine the dose-response based on cure rates of albendazole in preschool-aged children (2-5 years), school-aged children (6-12 years) and adults (≥ 21 years) infected with T. trichiura and hookworm.

The secondary objectives of the trial are to determine the efficacy based on egg reduction rates of albendazole in preschool-aged children, school-aged children and adults, to determine an exposure (including length of time that the drug concentration is above the MIC, Cmax, AUC)-response correlation of albendazole in preschool-aged children, school-aged children and adults, to evaluate the safety and tolerability of albendazole in preschool-aged children, school-aged children and adults, and to determine the efficacy against concomitant soil-transmitted helminthiasis (Ascaris lumbricoides).

After obtaining informed consent from individual/parents and/or caregiver, the medical history of the participants will be assessed with a standardized questionnaire, in addition to a clinical examination and venipuncture to examine biochemical parameters in the blood carried out by the study physician before treatment. Enrollment will be based on two stool samples that will be collected, if possible, on two consecutive days or otherwise within a maximum of 5 days.

All stool samples will be examined with duplicated Kato-Katz thick smears by experienced laboratory technicians. Randomization of participants into the treatment arms will be stratified according to intensity of infection. All participants will be interviewed before treatment, 3 and 24 hours and 3 weeks after treatment about the occurrence of adverse events. Children and adults will be sampled using finger pricking for micro-blood sampling at 0, 1, 2, 3, 4, 6, 8, 24 hours post-dosing.

The primary analysis will include all participants with primary end point data (available case analysis). Supplementary, a per-protocol analysis and an intention-to-treat analysis will be conducted. CRs will be calculated as the percentage of egg-positive subjects at baseline who become egg-negative after treatment. Differences among CRs will be analysed by using crude logistic regressions and adjusted logistic regressions (adjustment for age, sex, and height).

Geometric and arithmetic mean egg counts will be calculated for the different treatment arms before and after treatment to assess the corresponding ERRs. Bootstrap resampling method with 2,000 replicates will be used to calculate 95% confidence intervals (CIs) for differences in ERRs. Noncompartmental and nonlinear mixed-effects (NLME) modeling will be used to determine PK parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults (≥21 years), preschool-aged children (2-5 years) and school-aged children (6-12 years) infected with T. trichiura/hookworm
2. Written informed consent/assent signed from parent/guardian
3. Positive for T. trichiura/hookworm by at least two slides of the quadruple Kato-Katz thick smears and infection intensities of at least 100 eggs per gram of stool (EPG)
4. Agree to comply with study procedures, including provision of two stool samples at the beginning (baseline) and approximately three weeks after treatment (follow-up).

Exclusion Criteria:

1. Presence of acute or uncontrolled systemic illnesses (e.g. severe anemia, infection, clinical malaria) as assessed by a medical doctor, upon initial clinical assessment and liver function tests.
2. Known or reported history of chronic illness such as HIV, acute or chronic hepatitis, cancer, diabetes, chronic heart disease or renal disease.
3. Prior treatment with anthelmintics (eg, diethylcarbamazine [DEC], suramin, ivermectin, mebendazole or albendazole) within 4 weeks before planned test article administration.
4. Received any investigational drugs or investigational devices within 4 weeks before administration of test article that may confound safety and/or efficacy assessments.
5. Known or suspected allergy to benzimidazoles.
6. Pregnant (urine testing) or breastfeeding women

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Suisse de Recherches Scientifiques en Côte d'Ivoire (CSRS), Abidjan, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Patel C, Coulibaly JT, Hofmann D, N'Gbesso Y, Hattendorf J, Keiser J. Efficacy and Safety of Albendazole in Hookworm-infected Preschool-aged Children, School-aged Children, and Adults in Cote d'Ivoire: A Phase 2 Randomized, Controlled Dose-finding Trial. Clin Infect Dis. 2021 Jul 15;73(2):e494-e502. doi: 10.1093/cid/ciaa989. PMID 32668456
- [Derived] Patel C, Coulibaly JT, Schulz JD, N'Gbesso Y, Hattendorf J, Keiser J. Efficacy and safety of ascending dosages of albendazole against Trichuris trichiura in preschool-aged children, school-aged children and adults: A multi-cohort randomized controlled trial. EClinicalMedicine. 2020 May 5;22:100335. doi: 10.1016/j.eclinm.2020.100335. eCollection 2020 May. PMID 32405623

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Against T. Trichiura in PSAC: Placebo against T. trichiura in preschool-aged children
- ALB 200 mg Against T. Trichiura in PSAC: 200 mg of albendazole against T. trichiura in preschool-aged children
- ALB 400 mg Against T. Trichiura in PSAC: 400 mg of albendazole against T. trichiura in preschool-aged children
- ALB 600 mg Against T. Trichiura in PSAC: 600 mg of albendazole against T. trichiura in preschool-aged children
- Placebo Against T. Trichiura in SAC: Placebo against T. trichiura in school-aged children
- ALB 400 mg Against T. Trichiura in SAC: 400 mg of albendazole against T. trichiura in school-aged children
- ALB 600 mg Against T. Trichiura in SAC: 600 mg of albendazole against T. trichiura in school-aged children
- ALB 800 mg Against T. Trichiura in SAC: 800 mg of albendazole against T. trichiura in school-aged children
- Placebo Against T. Trichiura in Adults: Placebo against T. trichiura in adults
- ALB 400 mg Against T. Trichiura in Adults: 400 mg of albendazole against T. trichiura in adults
- ALB 600 mg Against T. Trichiura in Adults: 600 mg of albendazole against T. trichiura in adults
- ALB 800 mg Against T. Trichiura in Adults: 800 mg of albendazole against T. trichiura in adults
- Placebo Against Hookworm in PSAC: Placebo against hookworm in preschool-aged children
- ALB 200 mg Against Hookworm in PSAC: 200 mg of albendazole against hookworm in preschool-aged children
- ALB 400 mg Against Hookworm in PSAC: 400 mg of albendazole against hookworm in preschool-aged children
- ALB 600 mg Against Hookworm in PSAC: 600 mg of albendazole against hookworm in preschool-aged children
- Placebo Against Hookworm in SAC: Placebo against hookworm in school-aged children
- ALB 200 mg Against Hookworm in SAC: 200 mg of albendazole against hookworm in school-aged children
- ALB 400 mg Against Hookworm in SAC: 400 mg of albendazole against hookworm in school-aged children
- ALB 600 mg Against Hookworm in SAC: 600 mg of albendazole against hookworm in school-aged children
- ALB 800 mg Against Hookworm in SAC: 800 mg of albendazole against hookworm in school-aged children
- Placebo Against Hookworm in Adults: Placebo against hookworm in adults
- ALB 200 mg Against Hookworm in Adults: 200 mg of albendazole against hookworm in adults
- ALB 400 mg Against Hookworm in Adults: 400 mg of albendazole against hookworm in adults
- ALB 600 mg Against Hookworm in Adults: 600 mg of albendazole against hookworm in adults
- ALB 800 mg Against Hookworm in Adults: 800 mg of albendazole against hookworm in adults
Period: Overall Study
Arm/Group | Placebo Against T. Trichiura in PSAC | ALB 200 mg Against T. Trichiura in PSAC | ALB 400 mg Against T. Trichiura in PSAC | ALB 600 mg Against T. Trichiura in PSAC | Placebo Against T. Trichiura in SAC | ALB 400 mg Against T. Trichiura in SAC | ALB 600 mg Against T. Trichiura in SAC | ALB 800 mg Against T. Trichiura in SAC | Placebo Against T. Trichiura in Adults | ALB 400 mg Against T. Trichiura in Adults | ALB 600 mg Against T. Trichiura in Adults | ALB 800 mg Against T. Trichiura in Adults | Placebo Against Hookworm in PSAC | ALB 200 mg Against Hookworm in PSAC | ALB 400 mg Against Hookworm in PSAC | ALB 600 mg Against Hookworm in PSAC | Placebo Against Hookworm in SAC | ALB 200 mg Against Hookworm in SAC | ALB 400 mg Against Hookworm in SAC | ALB 600 mg Against Hookworm in SAC | ALB 800 mg Against Hookworm in SAC | Placebo Against Hookworm in Adults | ALB 200 mg Against Hookworm in Adults | ALB 400 mg Against Hookworm in Adults | ALB 600 mg Against Hookworm in Adults | ALB 800 mg Against Hookworm in Adults
Started | 27 | 27 | 30 | 27 | 46 | 45 | 46 | 43 | 10 | 11 | 9 | 12 | 0 (During screening, the principal investigator decided to remove the this arm due to recruitment.) | 13 | 13 | 12 | 24 | 27 | 27 | 29 | 26 | 40 | 41 | 38 | 40 | 37
Completed | 24 | 21 | 23 | 18 | 46 | 43 | 43 | 41 | 7 | 9 | 8 | 11 | 0 | 13 | 13 | 12 | 23 | 27 | 27 | 28 | 25 | 35 | 35 | 30 | 39 | 34
Not Completed | 3 | 6 | 7 | 9 | 0 | 2 | 3 | 2 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 5 | 6 | 8 | 1 | 3
Not completed — Lost to Follow-up | 3 | 6 | 7 | 9 | 0 | 2 | 3 | 2 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 5 | 6 | 8 | 1 | 3

BASELINE CHARACTERISTICS:
Population: The Placebo against hookworm in PSAC arm was removed from the trial after discussion with with principal investigators.
Groups:
- Placebo Against T. Trichiura in Adults: Placebo against T. trichiura in adults (>21 years)
- Placebo Against Hookworm in Adults: Placebo against hookworm in adults (>21 years)
- Total: Total of all reporting groups
Arm/Group | Placebo Against T. Trichiura in PSAC | ALB 200 mg Against T. Trichiura in PSAC | ALB 400 mg Against T. Trichiura in PSAC | ALB 600 mg Against T. Trichiura in PSAC | Placebo Against T. Trichiura in SAC | ALB 400 mg Against T. Trichiura in SAC | ALB 600 mg Against T. Trichiura in SAC | ALB 800 mg Against T. Trichiura in SAC | Placebo Against T. Trichiura in Adults | ALB 400 mg Against T. Trichiura in Adults | ALB 600 mg Against T. Trichiura in Adults | ALB 800 mg Against T. Trichiura in Adults | Placebo Against Hookworm in PSAC | ALB 200 mg Against Hookworm in PSAC | ALB 400 mg Against Hookworm in PSAC | ALB 600 mg Against Hookworm in PSAC | Placebo Against Hookworm in SAC | ALB 200 mg Against Hookworm in SAC | ALB 400 mg Against Hookworm in SAC | ALB 600 mg Against Hookworm in SAC | ALB 800 mg Against Hookworm in SAC | Placebo Against Hookworm in Adults | ALB 200 mg Against Hookworm in Adults | ALB 400 mg Against Hookworm in Adults | ALB 600 mg Against Hookworm in Adults | ALB 800 mg Against Hookworm in Adults | Total
Number analyzed (Participants) | 27 | 27 | 30 | 27 | 46 | 45 | 46 | 43 | 10 | 11 | 9 | 12 | 0 | 13 | 13 | 12 | 24 | 27 | 27 | 29 | 26 | 40 | 41 | 38 | 40 | 37 | 700
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 4.1 (0.9) | 4.0 (0.9) | 3.8 (1.1) | 4.0 (0.9) | 8.9 (1.9) | 8.9 (1.9) | 8.7 (2.0) | 8.8 (1.8) | 44.3 (12.3) | 40.5 (11.9) | 36.6 (12.2) | 44.8 (15.9) |  | 3.8 (1.2) | 3.8 (1.3) | 3.8 (1.1) | 9.1 (2.2) | 9.1 (1.9) | 9.8 (1.9) | 9.2 (2.2) | 9.4 (2.3) | 35.4 (10.3) | 39.8 (12.2) | 36.3 (12.2) | 39.2 (11.5) | 35.7 (12.0) | 17.7 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 16 | 18 | 25 | 15 | 19 | 17 | 6 | 9 | 7 | 8 |  | 5 | 9 | 8 | 8 | 12 | 8 | 5 | 7 | 7 | 16 | 7 | 7 | 9 | 282
  Male | 11 | 9 | 14 | 9 | 21 | 30 | 27 | 26 | 4 | 2 | 2 | 4 |  | 8 | 4 | 4 | 16 | 15 | 19 | 24 | 19 | 33 | 25 | 31 | 33 | 28 | 418
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
T. trichuris median eggs per gram [Median (Inter-Quartile Range); unit: eggs per gram of stool] | 216 [120 to 438] | 264 [96 to 558] | 210 [144 to 510] | 228 [150 to 726] | 387 [222 to 1068] | 426 [192 to 1266] | 507 [186 to 1134] | 414 [162 to 1116] | 138 [114 to 270] | 168 [114 to 504] | 156 [114 to 288] | 195 [150 to 402] |  | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 294 [162 to 972]
T. trichuris infection intensity [Count of Participants; unit: Participants]
  Light (1-999 epg) | 22 | 22 | 24 | 21 | 32 | 30 | 31 | 30 | 10 | 10 | 9 | 10 |  | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 260
  Moderate (1000-9999 epg) | 4 | 5 | 5 | 6 | 14 | 15 | 15 | 12 | 0 | 1 | 0 | 2 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 79
  Heavy (>= 10000 epg) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Not infected | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 13 | 13 | 11 | 22 | 25 | 27 | 29 | 24 | 39 | 41 | 38 | 40 | 36 | 358
hookworm median eggs per gram [Median (Inter-Quartile Range); unit: eggs per gram of stool] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] |  | 216 [150 to 618] | 126 [60 to 540] | 252 [111 to 423] | 183 [78 to 450] | 126 [72 to 336] | 138 [78 to 246] | 156 [84 to 528] | 153 [66 to 366] | 157 [96 to 318] | 126 [54 to 444] | 96 [54 to 264] | 189 [63 to 570] | 114 [84 to 216] | 132 [66 to 369]
hookworm infection intensity [Count of Participants; unit: Participants]
  Light (1-1999 epg) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 3 | 1 | 1 | 0 | 0 |  | 12 | 12 | 11 | 22 | 26 | 27 | 27 | 24 | 38 | 40 | 38 | 40 | 36 | 363
  Moderate (2000-3999 epg) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 1 | 1 | 1 | 2 | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 1 | 12
  Heavy (>= 4000 epg) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Not infected | 27 | 27 | 29 | 27 | 45 | 44 | 44 | 40 | 9 | 10 | 9 | 12 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 323
A. lumbricoides infection intensity [Count of Participants; unit: Participants]
  Light (1-4999 epg) | 2 | 2 | 3 | 2 | 8 | 8 | 4 | 6 | 0 | 1 | 0 | 2 |  | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 44
  Moderate (5000-49999 epg) | 2 | 6 | 2 | 1 | 5 | 9 | 6 | 7 | 0 | 2 | 0 | 1 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41
  Heavy (>= 50000 epg) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not infected | 23 | 19 | 25 | 24 | 33 | 27 | 36 | 30 | 10 | 8 | 9 | 9 |  | 12 | 13 | 11 | 23 | 26 | 27 | 28 | 26 | 40 | 41 | 38 | 39 | 37 | 614

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate Against T. Trichiura and Hookworm Infections
Description: The conversion from being egg positive pre-treatment to egg negative post-treatment, or cure rate (CR).
Time Frame: 14-21 days after treatment
Population: An analysis set of all randomized participants who provided any follow-up data was used to perform an available-case analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Against T. Trichiura in PSAC | ALB 200 mg Against T. Trichiura in PSAC | ALB 400 mg Against T. Trichiura in PSAC | ALB 600 mg Against T. Trichiura in PSAC | Placebo Against T. Trichiura in SAC | ALB 400 mg Against T. Trichiura in SAC | ALB 600 mg Against T. Trichiura in SAC | ALB 800 mg Against T. Trichiura in SAC | Placebo Against T. Trichiura in Adults | ALB 400 mg Against T. Trichiura in Adults | ALB 600 mg Against T. Trichiura in Adults | ALB 800 mg Against T. Trichiura in Adults | Placebo Against Hookworm in PSAC | ALB 200 mg Against Hookworm in PSAC | ALB 400 mg Against Hookworm in PSAC | ALB 600 mg Against Hookworm in PSAC | Placebo Against Hookworm in SAC | ALB 200 mg Against Hookworm in SAC | ALB 400 mg Against Hookworm in SAC | ALB 600 mg Against Hookworm in SAC | ALB 800 mg Against Hookworm in SAC | Placebo Against Hookworm in Adults | ALB 200 mg Against Hookworm in Adults | ALB 400 mg Against Hookworm in Adults | ALB 600 mg Against Hookworm in Adults | ALB 800 mg Against Hookworm in Adults
Number analyzed (Participants) | 24 | 21 | 23 | 18 | 46 | 43 | 43 | 41 | 7 | 9 | 8 | 11 | 0 | 13 | 13 | 12 | 23 | 27 | 27 | 28 | 25 | 35 | 35 | 30 | 39 | 34
Participants
  Cured | 4 | 2 | 4 | 5 | 3 | 7 | 11 | 7 | 1 | 5 | 4 | 3 |  | 9 | 8 | 10 | 10 | 17 | 20 | 18 | 19 | 5 | 16 | 16 | 22 | 32
  Not cured | 20 | 19 | 19 | 13 | 43 | 36 | 32 | 34 | 6 | 4 | 4 | 8 |  | 4 | 5 | 2 | 13 | 10 | 7 | 10 | 6 | 30 | 19 | 14 | 17 | 2

2. Secondary Outcome: Egg-reduction Rate (ERR) Against T. Trichiura and Hookworm Infections, Respectively
Description: Percent change in geometric mean eggs per gram of stool from before to after treatment
Time Frame: 14-21 days after treatment
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo Against T. Trichiura in PSAC | ALB 200 mg Against T. Trichiura in PSAC | ALB 400 mg Against T. Trichiura in PSAC | ALB 600 mg Against T. Trichiura in PSAC | Placebo Against T. Trichiura in SAC | ALB 400 mg Against T. Trichiura in SAC | ALB 600 mg Against T. Trichiura in SAC | ALB 800 mg Against T. Trichiura in SAC | Placebo Against T. Trichiura in Adults | ALB 400 mg Against T. Trichiura in Adults | ALB 600 mg Against T. Trichiura in Adults | ALB 800 mg Against T. Trichiura in Adults | Placebo Against Hookworm in PSAC | ALB 200 mg Against Hookworm in PSAC | ALB 400 mg Against Hookworm in PSAC | ALB 600 mg Against Hookworm in PSAC | Placebo Against Hookworm in SAC | ALB 200 mg Against Hookworm in SAC | ALB 400 mg Against Hookworm in SAC | ALB 600 mg Against Hookworm in SAC | ALB 800 mg Against Hookworm in SAC | Placebo Against Hookworm in Adults | ALB 200 mg Against Hookworm in Adults | ALB 400 mg Against Hookworm in Adults | ALB 600 mg Against Hookworm in Adults | ALB 800 mg Against Hookworm in Adults
Number analyzed (Participants) | 24 | 21 | 23 | 18 | 46 | 43 | 43 | 41 | 7 | 9 | 8 | 11 | 0 | 13 | 13 | 12 | 23 | 27 | 27 | 28 | 25 | 35 | 35 | 30 | 39 | 34
percent change | 79.1 [53.5 to 91.2] | 63.8 [33.1 to 83.1] | 87.1 [67.3 to 95.3] | 88.5 [70.4 to 95.7] | 55.9 [26.1 to 75.2] | 82.0 [67.8 to 90.5] | 88.4 [74.8 to 94.8] | 78.7 [60.5 to 89.1] | 85.2 [65.9 to 95.3] | 97.7 [86.7 to 99.8] | 94.7 [61.0 to 99.6] | 92.6 [71.9 to 98.5] |  | 99.0 [94.7 to 99.9] | 96.2 [83.5 to 99.4] | 99.6 [98.5 to 100.0] | 90.6 [72.3 to 97.3] | 97.7 [93.5 to 99.3] | 99.0 [97.4 to 99.7] | 98.3 [95.4 to 99.5] | 98.4 [95.9 to 99.6] | 33.0 [-27.1 to 67.3] | 93.8 [87.0 to 97.3] | 95.8 [90.2 to 98.3] | 97.0 [92.5 to 98.9] | 99.8 [99.5 to 100.0]

3. Secondary Outcome: Maximum Concentration (Cmax) of Albendazole Sulphoxide
Description: To determine maximum drug concentration (Cmax) of albendazole and its metabolites in adults (≥ 21 years), preschool-aged (2-5 years) and school-aged children (6-12 years). Albendazole sulfoxide will be quantified using a validated liquid chromatography tandem mass spectrometry (LC-MS/MS) method. Drug concentrations will be calculated by interpolation from a calibration curve with a foreseen limit of quantification of approximately 1-5 ng/ml.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 24 hours post-dosing
Measure: Mean (Standard Deviation); unit: mikromol/L
Arm/Group | ALB 200 mg Against T. Trichiura in PSAC | ALB 400 mg Against T. Trichiura in PSAC | ALB 600 mg Against T. Trichiura in PSAC | ALB 400 mg Against T. Trichiura in SAC | ALB 600 mg Against T. Trichiura in SAC | ALB 800 mg Against T. Trichiura in SAC | ALB 400 mg Against T. Trichiura in Adults | ALB 600 mg Against T. Trichiura in Adults | ALB 800 mg Against T. Trichiura in Adults | ALB 200 mg Against Hookworm in PSAC | ALB 400 mg Against Hookworm in PSAC | ALB 600 mg Against Hookworm in PSAC | ALB 200 mg Against Hookworm in SAC | ALB 400 mg Against Hookworm in SAC | ALB 600 mg Against Hookworm in SAC | ALB 800 mg Against Hookworm in SAC | ALB 200 mg Against Hookworm in Adults | ALB 400 mg Against Hookworm in Adults | ALB 600 mg Against Hookworm in Adults | ALB 800 mg Against Hookworm in Adults
Number analyzed (Participants) | 10 | 16 | 16 | 14 | 15 | 14 | 11 | 8 | 10 | 13 | 7 | 10 | 18 | 14 | 14 | 16 | 11 | 12 | 12 | 12
mikromol/L | 3.41 (2.58) | 6.61 (4.56) | 9.98 (7.16) | 3.67 (2.54) | 5.51 (3.778) | 7.14 (4.82) | 2.03 (1.44) | 2.95 (1.89) | 4.03 (2.62) | 1.70 (1.28) | 3.27 (2.28) | 4.98 (3.61) | 1.02 (0.74) | 2.11 (1.56) | 3.16 (2.41) | 4.12 (3.21) | 0.61 (0.44) | 1.22 (0.91) | 1.78 (1.20) | 2.43 (1.71)

4. Secondary Outcome: Time to Reach Cmax (Tmax) of Albendazole Sulphoxide
Description: To determine time to reach Cmax (tmax) of albendazole and its metabolites in adults (≥ 21 years), preschool-aged (2-5 years) and school-aged children (6-12 years). Albendazole sulfoxide was quantified using a validated liquid chromatography tandem mass spectrometry (LC-MS/MS) method. Drug concentrations will be calculated by interpolation from a calibration curve with a foreseen limit of quantification of approximately 1-5 ng/ml.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 24 hours post-dosing
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ALB 200 mg Against T. Trichiura in PSAC | ALB 400 mg Against T. Trichiura in PSAC | ALB 600 mg Against T. Trichiura in PSAC | ALB 400 mg Against T. Trichiura in SAC | ALB 600 mg Against T. Trichiura in SAC | ALB 800 mg Against T. Trichiura in SAC | ALB 400 mg Against T. Trichiura in Adults | ALB 600 mg Against T. Trichiura in Adults | ALB 800 mg Against T. Trichiura in Adults | ALB 200 mg Against Hookworm in PSAC | ALB 400 mg Against Hookworm in PSAC | ALB 600 mg Against Hookworm in PSAC | ALB 200 mg Against Hookworm in SAC | ALB 400 mg Against Hookworm in SAC | ALB 600 mg Against Hookworm in SAC | ALB 800 mg Against Hookworm in SAC | ALB 200 mg Against Hookworm in Adults | ALB 400 mg Against Hookworm in Adults | ALB 600 mg Against Hookworm in Adults | ALB 800 mg Against Hookworm in Adults
Number analyzed (Participants) | 10 | 16 | 16 | 14 | 15 | 14 | 11 | 8 | 10 | 13 | 7 | 10 | 18 | 14 | 14 | 16 | 11 | 12 | 12 | 12
hours | 6.8 (4.4) | 6.8 (3.8) | 6.8 (4.1) | 7.1 (4.6) | 7.0 (4.4) | 7.1 (4.3) | 7.3 (4.3) | 7.2 (4.3) | 7.4 (4.5) | 4.2 (2.7) | 4.2 (2.4) | 4.2 (2.6) | 4.5 (2.8) | 4.7 (3.1) | 4.7 (3.0) | 4.8 (3.0) | 5.3 (3.2) | 5.3 (3.2) | 5.4 (3.3) | 5.4 (3.4)

5. Secondary Outcome: Area Under the Curve (AUC) of Albendazole Sulphoxide
Description: To determine the area under the curve (AUC) of albendazole sulphoxide in adults (≥ 21 years), preschool-aged (2-5 years) and school-aged children (6-12 years). Albendazole and its metabolites (albendazole sulfoxide and albendazole sulfone) will be quantified using a validated liquid chromatography tandem mass spectrometry (LC-MS/MS) method. Drug concentrations will be calculated by interpolation from a calibration curve with a foreseen limit of quantification of approximately 1-5 ng/ml.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 24 hours post-dosing
Measure: Mean (Standard Deviation); unit: micogram/ml/h-1
Arm/Group | ALB 200 mg Against T. Trichiura in PSAC | ALB 400 mg Against T. Trichiura in PSAC | ALB 600 mg Against T. Trichiura in PSAC | ALB 400 mg Against T. Trichiura in SAC | ALB 600 mg Against T. Trichiura in SAC | ALB 800 mg Against T. Trichiura in SAC | ALB 400 mg Against T. Trichiura in Adults | ALB 600 mg Against T. Trichiura in Adults | ALB 800 mg Against T. Trichiura in Adults | ALB 200 mg Against Hookworm in PSAC | ALB 400 mg Against Hookworm in PSAC | ALB 600 mg Against Hookworm in PSAC | ALB 200 mg Against Hookworm in SAC | ALB 400 mg Against Hookworm in SAC | ALB 600 mg Against Hookworm in SAC | ALB 800 mg Against Hookworm in SAC | ALB 200 mg Against Hookworm in Adults | ALB 400 mg Against Hookworm in Adults | ALB 600 mg Against Hookworm in Adults | ALB 800 mg Against Hookworm in Adults
Number analyzed (Participants) | 10 | 16 | 16 | 14 | 15 | 14 | 11 | 8 | 10 | 13 | 7 | 10 | 18 | 14 | 14 | 16 | 11 | 12 | 12 | 12
micogram/ml/h-1 | 45.3 (31.4) | 90.3 (58.7) | 135.4 (89.6) | 47.3 (27.7) | 73.1 (44.2) | 96.9 (58.3) | 26.99 (15.9) | 40.2 (23.4) | 53.4 (29.9) | 16.6 (10.1) | 33.1 (18.8) | 49.5 (28.5) | 11.4 (6.7) | 22.3 (13.4) | 34.5 (22.1) | 45.2 (29.0) | 7.4 (4.0) | 14.9 (8.0) | 22.3 (12.1) | 29.8 (15.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at 3 hours and 24 hours after treatment.
Description: After a lengthy period of recruitment, it was decided to eliminate the placebo group for the PSAC cohort against hookworm.
Arm/Group | Placebo Against T. Trichiura in PSAC | ALB 200 mg Against T. Trichiura in PSAC | ALB 400 mg Against T. Trichiura in PSAC | ALB 600 mg Against T. Trichiura in PSAC | Placebo Against T. Trichiura in SAC | ALB 400 mg Against T. Trichiura in SAC | ALB 600 mg Against T. Trichiura in SAC | ALB 800 mg Against T. Trichiura in SAC | Placebo Against T. Trichiura in Adults | ALB 400 mg Against T. Trichiura in Adults | ALB 600 mg Against T. Trichiura in Adults | ALB 800 mg Against T. Trichiura in Adults | Placebo Against Hookworm in PSAC | ALB 200 mg Against Hookworm in PSAC | ALB 400 mg Against Hookworm in PSAC | ALB 600 mg Against Hookworm in PSAC | Placebo Against Hookworm in SAC | ALB 200 mg Against Hookworm in SAC | ALB 400 mg Against Hookworm in SAC | ALB 600 mg Against Hookworm in SAC | ALB 800 mg Against Hookworm in SAC | Placebo Against Hookworm in Adults | ALB 200 mg Against Hookworm in Adults | ALB 400 mg Against Hookworm in Adults | ALB 600 mg Against Hookworm in Adults | ALB 800 mg Against Hookworm in Adults
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/30 | 0/27 | 0/46 | 0/45 | 0/46 | 0/43 | 0/10 | 0/11 | 0/9 | 0/12 | 0/0 | 0/13 | 0/13 | 0/12 | 0/24 | 0/27 | 0/27 | 0/29 | 0/26 | 0/40 | 0/41 | 0/38 | 0/40 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/27 | 0/30 | 0/27 | 0/46 | 0/45 | 0/46 | 0/43 | 0/10 | 0/11 | 0/9 | 0/12 | 0/0 | 0/13 | 0/13 | 0/12 | 0/24 | 0/27 | 0/27 | 0/29 | 0/26 | 0/40 | 0/41 | 0/38 | 0/40 | 0/37
Other Adverse Events (participants affected / at risk) | 3/27 | 2/27 | 3/30 | 2/27 | 4/46 | 9/45 | 8/46 | 8/43 | 3/10 | 3/11 | 2/9 | 2/12 | 0/0 | 1/13 | 0/13 | 1/12 | 2/24 | 3/27 | 2/27 | 1/29 | 3/26 | 2/40 | 4/41 | 5/38 | 3/40 | 4/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Against T. Trichiura in PSAC (N=27) | ALB 200 mg Against T. Trichiura in PSAC (N=27) | ALB 400 mg Against T. Trichiura in PSAC (N=30) | ALB 600 mg Against T. Trichiura in PSAC (N=27) | Placebo Against T. Trichiura in SAC (N=46) | ALB 400 mg Against T. Trichiura in SAC (N=45) | ALB 600 mg Against T. Trichiura in SAC (N=46) | ALB 800 mg Against T. Trichiura in SAC (N=43) | Placebo Against T. Trichiura in Adults (N=10) | ALB 400 mg Against T. Trichiura in Adults (N=11) | ALB 600 mg Against T. Trichiura in Adults (N=9) | ALB 800 mg Against T. Trichiura in Adults (N=12) | Placebo Against Hookworm in PSAC (N=0) | ALB 200 mg Against Hookworm in PSAC (N=13) | ALB 400 mg Against Hookworm in PSAC (N=13) | ALB 600 mg Against Hookworm in PSAC (N=12) | Placebo Against Hookworm in SAC (N=24) | ALB 200 mg Against Hookworm in SAC (N=27) | ALB 400 mg Against Hookworm in SAC (N=27) | ALB 600 mg Against Hookworm in SAC (N=29) | ALB 800 mg Against Hookworm in SAC (N=26) | Placebo Against Hookworm in Adults (N=40) | ALB 200 mg Against Hookworm in Adults (N=41) | ALB 400 mg Against Hookworm in Adults (N=38) | ALB 600 mg Against Hookworm in Adults (N=40) | ALB 800 mg Against Hookworm in Adults (N=37)
Inpatient hospitalization due to clinical malaria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Against T. Trichiura in PSAC (N=27) | ALB 200 mg Against T. Trichiura in PSAC (N=27) | ALB 400 mg Against T. Trichiura in PSAC (N=30) | ALB 600 mg Against T. Trichiura in PSAC (N=27) | Placebo Against T. Trichiura in SAC (N=46) | ALB 400 mg Against T. Trichiura in SAC (N=45) | ALB 600 mg Against T. Trichiura in SAC (N=46) | ALB 800 mg Against T. Trichiura in SAC (N=43) | Placebo Against T. Trichiura in Adults (N=10) | ALB 400 mg Against T. Trichiura in Adults (N=11) | ALB 600 mg Against T. Trichiura in Adults (N=9) | ALB 800 mg Against T. Trichiura in Adults (N=12) | Placebo Against Hookworm in PSAC (N=0) | ALB 200 mg Against Hookworm in PSAC (N=13) | ALB 400 mg Against Hookworm in PSAC (N=13) | ALB 600 mg Against Hookworm in PSAC (N=12) | Placebo Against Hookworm in SAC (N=24) | ALB 200 mg Against Hookworm in SAC (N=27) | ALB 400 mg Against Hookworm in SAC (N=27) | ALB 600 mg Against Hookworm in SAC (N=29) | ALB 800 mg Against Hookworm in SAC (N=26) | Placebo Against Hookworm in Adults (N=40) | ALB 200 mg Against Hookworm in Adults (N=41) | ALB 400 mg Against Hookworm in Adults (N=38) | ALB 600 mg Against Hookworm in Adults (N=40) | ALB 800 mg Against Hookworm in Adults (N=37)
Headache (Nervous system disorders) | 1 | 2 | 3 | 0 | 3 | 1 | 3 | 5 | 1 | 3 | 2 | 2 | NA | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 3 | 4 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 4 | 4 | 3 | 7 | 2 | 3 | 1 | 0 | NA | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 3 | 0 | 1 | 1 | 2 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Infections and infestations) | 1 | 0 | 2 | 1 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT03527745/Prot_SAP_000.pdf